CLINICAL TRIAL: NCT04268173
Title: Community-Based, Client-Centered Prevention Homes to Address the Rural Opioid Epidemic- Aim 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Tulane University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-0866; UH3DA044826 (NIH); A534265 (Other: UW Madison); SMPH/MEDICINE/INFECT DIS (Other: UW Madison); Protocol Version 2/1/2023 (Other: UW Madison)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Drug Use Disorders; Hepatitis C; Harm Reduction; Opioid-use Disorder
MeSH Terms: conditions — Substance-Related Disorders; Hepatitis C; Harm Reduction; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants were enrolled in a 2-arm, non-randomized intervention trial based on the location where they received harm reduction services. Harm reduction clients receiving services at offices in 3 selected Wisconsin counties (La Crosse, Brown, and Marathon) were assigned to work with a Prevention Navigator at the office location, while clients receiving services in other counties (Douglas, Eau Claire, and Outagamie) received usual services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention Navigation (Experimental): Participants enrolled in this arm will receive a 12-week community-based, client-centered, prevention intervention.
  Interventions: Other: Community-Based, Client-Centered Prevention Home
- Usual Services (No Intervention): Participants enrolled in this arm will receive services as usual from Vivent Health and will not engage in the intervention.

INTERVENTIONS:
Other: Community-Based, Client-Centered Prevention Home — Prevention Navigators at Vivent Helath offices will engage participants in risk assessments, goal planning, and treatment referrals based on their needs and desires.
  Other Names: Prevention Navigation
  Arms: Prevention Navigation

SUMMARY:
The goal of this study was to effectively use a client-centered community-based intervention to engage people who inject drugs (PWIDs) in healthcare that helps reduce risky behaviors and lower infectious disease risks. Participants in the intervention group of this study received a 12-week intensive multilevel harm reduction case-management intervention at three rural Vivent Health offices. Service coordination aimed to reduce human immunodeficiency virus (HIV), hepatitis C virus (HCV), and overdose risks in PWIDs. Prevention Navigators (PNs) at each office helped to coordinate referrals to reduce substance use disorder and increase engagement in the substance use disorder care cascades.

DETAILED DESCRIPTION:
This project was conducted by an experienced, interdisciplinary team working across academic, public health, and non-government sectors. The main community partner Vivent Health, formerly known as the AIDS Resource Center of Wisconsin (ARCW), is a unique, state-wide organization that provides harm reduction services, including syringe services and confidential HIV and HCV testing, to clients at 10 fixed sites and numerous mobile units reaching all 72 Wisconsin counties. Based on the investigators' preliminary studies and prior collaborations, the investigators selected 6 counties in rural Wisconsin. The Client-Centered Prevention Home intervention model was implemented at 3 Vivent Health field offices in 3 of these counties, and 3 other counties served as "usual services," or control sites. Participants in the intervention underwent a 12-week intensive multilevel harm reduction case-management intervention geared towards coordinating referrals to reduce substance use disorder and increase engagement in the substance use disorder care cascades, and reduce vulnerability to HIV, STIs, and HCV and increase in engagement in the HIV, STI, and HCV care cascades. Participants in the intervention arm worked with Prevention Navigators to undergo a risk assessment and identify problems and create goals that they want to achieve. Each session after that was used to review the needs assessment and goals. During their last meeting, participants and prevention navigators developed a discharge plan that will enable the participants to work on their goals on their own. Participants at all six sites were offered rapid testing for HIV, HCV, and STIs, and fill out survey questionnaires to evaluate risk behaviors, intervention effectiveness, and general needs of the communities.

ELIGIBILITY:
Inclusion Criteria:

* has injected drugs in the past 30 days, resides in Wisconsin, over 18 years of age
* able to read and write in English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Westergaard, MD, PhD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - Vivent Health, Appleton, Wisconsin
  - Vivent Health, Eau Claire, Wisconsin
  - Vivent Health, Green Bay, Wisconsin
  - Vivent Health, La Crosse, Wisconsin
  - Vivent Health, Schofield, Wisconsin
  - Vivent Health, Superior, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification. Proposals should be directed to the Data coordinating center at University of Washington. If approved after review, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after upload to the data coordinating center at University of Washington and will remain for the time records must be held for, according to our data use agreement.
Access Criteria: Data will only be shared among researchers in the cooperative agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 343 individuals enrolled in the study and provided informed consent. Of these, 16 withdrew from the study or were lost to follow-up before participating in any data collection. Results are therefore reported only for N=327 who completed at least a baseline study assessment.
Period: Overall Study
Arm/Group | Usual Services | Prevention Navigation
Started | 133 | 194
Completed | 58 | 86
Not Completed | 75 | 108
Not completed — Lost to Follow-up | 75 | 108

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Services | Prevention Navigation | Total
Number analyzed (Participants) | 133 | 194 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.1) | 38.2 (10.0) | 38.2 (10.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 49 | 84 | 133
  Male | 83 | 107 | 190
  Other | 1 | 2 | 3
  Unknown | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 13 | 17
  Not Hispanic or Latino | 128 | 180 | 308
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 22 | 27
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 121 | 154 | 275
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 133 | 194 | 327

OUTCOME MEASURES:

1. Primary Outcome: Change in the Addiction Treatment Accessibility and Utilization as Assessed by Change in Likert Scale
Description: The following question was asked on a scale of 0 to 4, where 0=strongly disagree and 4=strongly agree:
  If I wanted to start medical treatment for opioid or heroin addiction, I could easily get buprenorphine or Suboxone or Subutex.
  The outcome is represented as the mean response in each intervention group (min 0, max 4)
Time Frame: Pre-intervention, post intervention (3 months)
Population: Participants responding to the survey question were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Services | Prevention Navigation
Number analyzed (Participants) | 103 | 148
score on a scale
  Pre-intervention | 1.26 (1.10) | 1.07 (1.21)
  Post-intervention: number analyzed (Participants) | 50 | 148
  Post-intervention | 1.12 (1.15) | 1.03 (1.30)
Statistical Analysis 1: Comparison: Prevention Navigation; Test type: Equivalence — A two sample t-test was conducted to test the null hypothesis that the pre-intervention mean response was equivalent to the post-intervention mean response in the Prevention Navigation group. Hypothesis: A p-value greater than 0.05 suggests the means are not statistically different from one another; p = 0.84, t-test, 2 sided

2. Primary Outcome: Change in the Addiction Treatment Accessibility and Utilization as Assessed by Change in Frequency of "Yes" Answers
Description: Following questions will be asked with yes or no answers.
  In the past 3 months, have you gotten buprenorphine maintenance medication-like Suboxone or Subutex-from a doctor or program? Responses were coded as 0 = "No" and 1 = "Yes." Summary statistics presented as "mean" below represent the proportion responding yes.
Time Frame: Pre-intervention, post intervention (3 months)
Population: Only participants responding to the survey question were analyzed
Measure: Mean (Standard Deviation); unit: proportion of "Yes" responses
Arm/Group | Usual Services | Prevention Navigation
Number analyzed (Participants) | 132 | 185
proportion of "Yes" responses
  Pre-Intervention | 0.17 (0.38) | 0.16 (0.37)
  Post-Intervention: number analyzed (Participants) | 54 | 83
  Post-Intervention | 0.037 (0.19) | 0.11 (0.31)

3. Primary Outcome: Change in the Risk of HIV as Assessed by Change in Likert Scale
Description: Following questions will be asked to gauge ease of accessing clean injecting equipment to assess how risky the participants behaviors are in relation to HIV transmission.
  "It's easy for me to get new, clean syringes or needles."
  Questions will be answered on a scale of 0 to 4, with 0=strongly disagree and 4=strongly agree. An increase in the Likert scale among intervention participants is associated with increased access to HIV prevention compared to the controls.
Time Frame: Pre-intervention, post intervention (3 months)
Population: Only participants responding to the survey question were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Services | Prevention Navigation
Number analyzed (Participants) | 112 | 135
score on a scale
  Pre-intervention | 1.05 (1.01) | 1.09 (1.05)
  Post-intervention: number analyzed (Participants) | 46 | 135
  Post-intervention | 1.28 (1.04) | 0.86 (1.17)

4. Primary Outcome: Change in the Risk of HIV as Assessed by Risky Behavior Frequencies
Description: Participants were asked to gauge frequency of safe injection behaviors that reduce the risk of HIV. Participants will be asked how many times in the last 30 days they have practiced these behaviors.
  "In the last 3 months, how often have you shared needles with someone else, used a syringe more than once, used equipment you knew wasn't clean, or received equipment from a potentially unsafe source?"
  Responses were coded 0="never" and 1="at least once"
Time Frame: Pre-intervention, post intervention (3 months)
Population: Participants who responded to the survey question were analyzed
Measure: Mean (Standard Deviation); unit: proportion reporting "at least once"
Arm/Group | Usual Services | Prevention Navigation
Number analyzed (Participants) | 131 | 190
proportion reporting "at least once"
  Pre-intervention | 0.24 (0.43) | 0.25 (0.44)
  Post-intervention: number analyzed (Participants) | 58 | 85
  Post-intervention | 0.19 (0.40) | 0.21 (0.41)

5. Primary Outcome: Change in the Risk of Drug Overdose as Assessed by Change in Likert Scale
Description: Following question will be asked on a scale of 0 to 4, where 0=strongly disagree and 4=strongly agree
  "If I wanted the overdose reversal drug naloxone or Narcan, I could easily get it."
Time Frame: Pre-intervention, post intervention (3 months)
Population: Participants responding to the survey question were analyzed
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Services | Prevention Navigation
Number analyzed (Participants) | 126 | 180
score on a scale
  Pre-intervention | 0.52 (0.82) | 0.42 (0.85)
  Post-intervention: number analyzed (Participants) | 53 | 80
  Post-intervention | 0.57 (1.01) | 0.56 (1.17)

6. Other Pre Specified Outcome: Change in the Risk of Viral Hepatitis as Assessed by Change in Likert Scale
Time Frame: Baseline, 3 months, and 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Smoking Frequency as Assessed by Self-reported Behaviors
Time Frame: Baseline, 3 months, and 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Self-stigma as Assessed by Change in Likert Scale
Time Frame: Baseline, 3 months, and 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in the Risk of Drug Overdose as Assessed by Change in Frequency of Narcan Distribution
Time Frame: Baseline, 3 months, and 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in the Treatment Frequency of Viral Hepatitis as Assessed by Wisconsin(WI) Surveillance Databases and Medicaid Data
Time Frame: Baseline, 3 months, and 6 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Addiction Treatment Accessibility and Utilization Frequency Assessment From Long Term Medicaid Data
Time Frame: Year 2
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Hepatitis C Treatment Frequency From Long Term Medicaid Data
Time Frame: Year 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The time period during which participants were observed lasted from the date of enrollment until completion of the final follow-up survey (approximately 3-6 months).
Description: Because this is a minimal risk study, in which procedures were limited to collection of survey data, the frequency of specific adverse events were not systematically collected. If the study team became aware of a participant hospitalization or death, however, information about the event would be recorded and shared with the institutional review board.
Arm/Group | Usual Services | Prevention Navigation
All-Cause Mortality (participants affected / at risk) | 0/133 | 2/194
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/194
Other Adverse Events (participants affected / at risk) | 0/133 | 0/194

LIMITATIONS AND CAVEATS:
This trial was conducted in a challenging community setting among a vulnerable population affected by severe substance use disorder, unstable housing, and frequent criminal legal system involvement. As a result, we experienced very high levels of attrition in both study arms. The resulting level of missing data significantly impedes the ability to draw conclusions about the relationship between intervention exposure and any of the study outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT04268173/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT04268173/ICF_001.pdf